CLINICAL TRIAL: NCT07160244
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blinded Trial to Evaluate the Safety, Tolerability, and Immunogenicity of a Multivalent Group B Streptococcus Vaccine in Healthy Pregnant Women and Their Infants
Brief Title: BEATRIX: A Study to Learn About a Group B Streptococcus Vaccine in Healthy Pregnant Women and Their Babies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C1091009; 2022-503070-36-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-08-14; First posted 2025-09-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: group B streptococcus, maternal immunization, vaccine
MeSH Terms: interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PEDIARIX; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- GBS6 (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- Infanrix hexa (Experimental): Commercially available combination vaccine containing diphtheria, tetanus, pertussis (whooping cough), hepatitis B, poliomyelitis (polio), and Haemophilus influenzae type b (Hib)
  Interventions: Biological: Infanrix hexa
- Prevenar 20 (Experimental): Commercially available vaccine that protects against 20 strains of Streptococcus pneumoniae
  Interventions: Biological: Prevenar 20
- Pediarix (Experimental): Commercially available combination vaccine containing diphtheria, tetanus, pertussis (whooping cough), hepatitis B, and polio
  Interventions: Biological: Pediarix
- Prevnar 20 (Experimental): Commercially available vaccine that protects against 20 strains of Streptococcus pneumoniae
  Interventions: Biological: Prevnar 20
- Infanrix (Experimental): Commercially available combination vaccine containing diphtheria, tetanus, and pertussis
  Interventions: Biological: Infanrix

INTERVENTIONS:
Biological: Multivalent Group B streptococcus vaccine — Multivalent Group B streptococcus vaccine
  Other Names: GBS6
  Arms: GBS6
Biological: Placebo — Saline Control
  Arms: Placebo
Biological: Infanrix hexa — Vaccine administered in a subset of infant participants as per the national immunization schedule
  Arms: Infanrix hexa
Biological: Prevenar 20 — Vaccine administered in a subset of infant participants as per the national immunization schedule
  Arms: Prevenar 20
Biological: Pediarix — Vaccine administered in a subset of infant participants as per the national immunization schedule
  Arms: Pediarix
Biological: Prevnar 20 — Vaccine administered in a subset of infant participants as per the national immunization schedule
  Arms: Prevnar 20
Biological: Infanrix — Vaccine administered in a subset of infant participants as per the national immunization schedule
  Arms: Infanrix

SUMMARY:
BEATRIX (group B strEptococcus mATeRnal and Infant VaX study) The purpose of this study is to learn about the safety and how the group B streptococcus (GBS) vaccine works in pregnant women and their babies.

This study is seeking healthy pregnant participants:

* aged 49 or younger who can join.
* between 24 and 36 weeks of gestation ("Gestational age" is a medical term used to describe how far along your pregnancy is)
* had a fetal ultrasound examination performed with no major fetal abnormalities observed
* documented negative for HIV, syphilis and Hepatitis B All participants in this study will receive only 1 shot in an arm. This could either be a group B streptococcus 6-valent polysaccharide conjugate vaccine (GBS6) or placebo. Placebo is an inactive substance used in the study for comparison purposes; in this study, the placebo injection will be saline (saltwater). The pregnant participants may take part in this study for a maximum of 14 months (6 months after delivery) , and their babies for about 12 months after they are born. The pregnant participants will need to visit the research site at least 3 to 4 times with some visits permitted to occur over the telephone.

A subset of infants will be asked to take part in the study for up to 19 months. The subset will receive diphtheria toxoid-containing vaccine and/or pneumococcal vaccine following each country's standard immunization plan and have blood drawn 1 month after completion of the primary and/or toddler (booster) doses.

ELIGIBILITY:
Key Inclusion criteria- Maternal:

* Healthy pregnant women ≤49 years of age who are between 24 0/7 and 36 0/7 weeks of gestation on the day of planned vaccination, with an uncomplicated, singleton pregnancy, and who have no known increased risk of complications.
* Had a fetal anomaly ultrasound examination with no significant fetal abnormalities observed.
* Documented negative human immunodeficiency virus (HIV) antibody test, syphilis test, and hepatitis B virus (HBV) surface antigen test during this pregnancy and prior to randomization.
* Capable of giving personal signed informed consent.
* Willing to give informed consent for her infant to participate in the study.

Key Exclusion criteria- Maternal:

* Prepregnancy body mass index (BMI) of >40 kg/m2.
* Current pregnancy complications or abnormalities that may increase the risk associated with the participation in and completion of the study.
* Prior pregnancy complications or abnormalities that, based on the investigator's judgment, may increase the risk associated with the participation in and completion of the study.
* History of microbiologically proven invasive disease caused by GBS in the current pregnancy.
* A known or suspected infection during the current pregnancy that may increase the risk of complications in pregnancy (eg, active tuberculosis, syphilis, primary genital herpes simplex, malaria).

Key Inclusion criteria- Infant Participants

- Evidence of a signed and dated ICD signed by the parent(s)/legally authorized representative or legal guardian

Key Exclusion Criteria - Infant Participants:

- Children or grandchildren who are direct descendants of investigator site staff or sponsor and sponsor delegate employees directly involved in the conduct of the study.

Key Exclusion Criteria - Infant immunogenicity subset Participants:

- Children with a known or suspected contraindication to any vaccine administered in the infant vaccine immunogenicity subset.

Refer to the study contact for further eligibility details

Ages: 1 Day to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-11-06 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of maternal participants reporting prespecified local reactions within 7 days following study intervention | Within 7 days
The proportion of maternal participants reporting prespecified systemic events within 7 days following study intervention | Within 7 days
The proportion of maternal participants reporting adverse events (AEs) through 1 month following study intervention | 1 month
The proportion of maternal participants reporting serious adverse events (SAEs) through 6 months after delivery | 6 months after delivery
The proportion of maternal participants reporting medically attended adverse events (MAAEs) through 6 months after delivery | 6 months after delivery
The proportion of infant participants born to pregnant women who were vaccinated with GBS6 during pregnancy reporting adverse events (AEs) from birth through 1 month of age | Birth to 1 month of age
The proportion of infant participants born to pregnant women who were vaccinated with GBS6 during pregnancy reporting serious adverse events (SAEs) from birth through end of the study | Through study completion, at least 1 year
The proportion of infant participants born to pregnant women who were vaccinated with GBS6 during pregnancy reporting medically attended events (MAAEs) from birth through 6 months of age | Birth to 6 months of age
To measure the relative risk reduction in the proportion of infant participants at birth with GBS serotype-specific IgG antibody concentrations below predefined serotype-specific GBS late onset disease thresholds in the GBS6 group to the placebo group | Birth
To measure the relative risk reduction in the proportion of infant participants at birth with GBS serotype-specific IgG antibody concentrations below predefined serotype-specific GBS early onset disease thresholds in the GBS6 group to the placebo group | Birth
To evaluate the aggregate predicted VE combining all 6 serotypes in GBS6 to provide protection from invasive GBS late onset disease based on serotype specific anti-CPS IgG concentrations measured in infants at birth. | Birth
To evaluate the aggregate predicted VE combining all 6 serotypes in GBS6 to provide protection from invasive GBS early onset disease based on serotype specific anti-CPS IgG concentrations measured in infants at birth. | Birth

SECONDARY OUTCOMES:
To measure GBS serotype-specific opsonophagocytic titers in infant participants at birth by geometric mean ratio between GBS6 group versus placebo group and by the difference in seroresponse rates between GBS6 group and placebo group | Birth
To describe anti-CPS IgG antibody levels predicted to provide protection from invasive GBS disease (all disease) caused by the 6 individual vaccine serotypes in infants when GBS6 is administered to healthy pregnant women. | Birth
To describe anti-CPS IgG antibody levels in infant participants born to maternal participants vaccinated with GBS6. | Birth
To describe anti-CPS IgG antibody levels predicted to provide protection from invasive GBS LOD and EOD, separately, caused by the 6 individual vaccine serotypes (Ia, Ib, II, III, IV, and V) in infants when GBS6 is administered to healthy pregnant women. | Birth
To measure GBS serotype-specific IgG by geometric mean concentration in maternal participants at 1 month after vaccination and at delivery. | 1 month after vaccination and at delivery
Compare the proportion of infants with anti-diphtheria toxoid and pneumococcal IgG responses at 1 month post-primary and toddler doses between GBS6 and placebo groups, including predefined IgG levels and geometric mean ratios. | 1 month after the primary vaccination series and 1 month after the toddler dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (103):
- United States (54):
  - SEC Clinical Research, Dothan, Alabama
  - ClinMed, Phoenix, Arizona
  - Genesis OB/GYN, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Antelope Valley Medical Center, Lancaster, California
  - Chemidox Clinical Trials, Lancaster, California
  - South Florida Clinical Research Institute - Margate, Margate, Florida
  - Citadelle Clinical Research, North Miami Beach, Florida
  - Emerald Coast OBGYN Clinical Research, Panama City, Florida
  - HCA Florida Gulf Coast Hospital, Panama City, Florida
  - Advanced Specialty Research, Boise, Idaho
  - Express Lab, Garden City, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - Madison Memorial Hospital, Rexburg, Idaho
  - Accellacare - McFarland, Ames, Iowa
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic, PC, Ames, Iowa
  - Velocity Clinical Research, Covington, Covington, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Boeson Research GTF, Great Falls, Montana
  - Origin Health GTF, Great Falls, Montana
  - Boeson Research MSO, Missoula, Montana
  - Origin Health, Missoula, Montana
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Midwest Children's Health Research Center, Lincoln, Nebraska
  - Bryan Health, Lincoln, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Women's Health Care Center of Williamsburg, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Stony Brook Medicine Clinical Research Center, East Setauket, New York
  - ACGC Research, NYU Ambulatory Care Garden City, Garden City, New York
  - NYU Langone Ambulatory Care Garden City, Garden City, New York
  - NYU Langone Long Island, Clinical Research Center 3-002 (Admin only), Mineola, New York
  - Stony Brook University, Stony Brook, New York
  - Tribe Clinical Research, LLC- Greer, Greer, South Carolina
  - Tribe Clinical Research at Parkside Pediatrics Five Forks, Simpsonville, South Carolina
  - Proactive Clinical Research LLC, Edinburg, Texas
  - Memorial Hermann Memorial City Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Maximos Ob/Gyn, League City, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - The Group For Women - Kempsville Office, Norfolk, Virginia
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Womens Care Center, Norfolk, Virginia
  - Virginia Physicians For Women (VPFW), North Chesterfield, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Seattle Childrens Research Institute, Seattle, Washington
  - Seattle Childrens Hospital, Seattle, Washington
  - UW Medical Center Northwest, Seattle, Washington
  - UW Medical Center Montlake, Seattle, Washington
- Argentina (4):
  - Fundación Respirar, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Instituto de Maternidad y Ginecología Nuestra Señora de las Mercedes, San Miguel de Tucumán, Tucumán Province
  - Equipo Ciencia, Buenos Aires
- Finland (6):
  - FVR, Kokkolan rokotetutkimusklinikka, Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka, Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka, Tampere, Pirkanmaa
  - FVR, Seinäjoen rokotetutkimusklinikka, Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka, Turku, Southwest Finland
  - MeVac - Meilahti Vaccine Research Center, Helsinki, Uusimaa
- Japan (9):
  - St.Mary's Hospital, Kurume, Fukuoka
  - Sendai City Hospital, Sendai, Miyagi
  - Beppu Medical Center, Beppu-shi, Oita Prefecture
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Taniguchi Hospital, Izumisano, Osaka
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukui Aiiku Hospital, Fukui
  - Rakuwakai Otowa Hospital, Kyoto
  - Shizuoka General Hospital, Shizuoka
- South Korea (4):
  - Chonnam National University Hospital, Gwangju, Kwangju-kwangyǒkshi
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-kwangyǒkshi
  - Kyung Hee University Hospital at Gangdong, Seoul
- Spain (6):
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario HM Puerta del Sur, Madrid, Madrid, Comunidad de
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Antequera, Antequera
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (5):
  - Hsinchu Municipal Mackay Children's Hospital, Hsinchu, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (15):
  - University Hospitals Bristol NHS Foundation Trust, Bristol, Bristol, CITY of
  - St Michael's Hospital, Bristol, Bristol, CITY of
  - Barnet Hospital, London, England
  - St. George's Hospital, London, England
  - North Manchester General Hospital, Manchester, England
  - The Royal Cornwall Hospital, Truro, England
  - Southampton General Hospital, Southampton, Hampshire
  - St Mary's Hospital (Manchester University NHS Foundation Trust), Manchester, Lancashire
  - Imperial College Healthcare NHS Foundation Trust - St Mary's Hospital, London, London, CITY of
  - The Princess Royal Hospital, Shropshire, Telford AND Wrekin
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Royal Infirmary, Bristol
  - St James's University Hospital, Leeds
  - Royal Free Hospital, London
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1091009